CLINICAL TRIAL: NCT02097940
Title: Influence of Sensorimotor Treatment in the Balance of Soccer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Christiane Macedo, Doctor, Universidade Estadual de Londrina
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Christiane Macedo
Record Dates: First submitted 2014-03-17; First posted 2014-03-27 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Ankle Sprain
Keywords: Postural balance; Athletes; Sports; Soccer; Physiotherapy
MeSH Terms: conditions — Ankle Injuries | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment (Active Comparator): The treatment group performed of proprioceptive exercises with shifts and one-leg jumps.
  Interventions: Other: proprioceptive exercises
- control (No Intervention): The control group remained in soccer training

INTERVENTIONS:
Other: proprioceptive exercises — Exercises with movements, jumping and imbalance.
  Other Names: treatment
  Arms: treatment

SUMMARY:
This study presents the hypothesis that the sensory processing engine improves balance and agility for football athletes.

DETAILED DESCRIPTION:
Objectives: To investigate the influence of the sensorimotor treatment in balance, agility and functionality soccer players assessed using force platform, functional tests and questionnaires.

Methods: This study was characterized as a randomized clinical trial. 20 male soccer players was assessed by means of questionnaires, force platform in one foot, and functional tests of balance and agility (Side Hop Test, Figure of Eight Hop Star Excursion Balance Test and Test). To the platform, the parameters of the center pressure (COP) in the anterior- posterior and medial -lateral directions was used for analysis, to functional tests the time-second performance was analyzed. Initially all athletes respond to the questionnaires, was evaluated on the force platform and through functional testing by blind evaluators. Following, they were randomized to treatment groups (n=10) and control (n=10). The treatment group performed 6 weeks of proprioceptive exercises with shifts and one-leg jumps and bipedal support.

The control group remained in soccer training. At the end of the treatment protocol and all were reassessed following the cross-over, where the control group performed the same treatment sensory motor was developed.

ELIGIBILITY:
Inclusion Criteria:

* minimum of three years of training in the sport,
* participating in state and national competitions,
* often training at least five times a week

Exclusion Criteria:

* athletes undergoing surgical procedures or have muscle and joint injuries in the lower limbs in the last three months,
* which are in physical therapy or who require the use of stabilizers to perform the tests on the platform or during the treatment protocol

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
answers to survey | up to one year
  The athletes answered questionnaires with general data (age, weight, height, BMI, playing position)

SECONDARY OUTCOMES:
Variables center pressure swing | up to one year
  Evaluation of body balance on the force platform.

OTHER OUTCOMES:
time to perform the test | up to one year
  Functional tests have been developed (Side Hop Test, Figure of Eight Hop Star Excursion Balance Test and Test)

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Macedo, doctor, Principal Investigator — State University of Londrina
Locations (1):
- Junior Football Team, Londrina, Paraná, Brazil

REFERENCES:
- [Result] Emery CA, Meeuwisse WH. The effectiveness of a neuromuscular prevention strategy to reduce injuries in youth soccer: a cluster-randomised controlled trial. Br J Sports Med. 2010 Jun;44(8):555-62. doi: 10.1136/bjsm.2010.074377. PMID 20547668
- [Result] Bizzini M, Junge A, Dvorak J. Implementation of the FIFA 11+ football warm up program: how to approach and convince the Football associations to invest in prevention. Br J Sports Med. 2013 Aug;47(12):803-6. doi: 10.1136/bjsports-2012-092124. Epub 2013 Jun 27. PMID 23813485